CLINICAL TRIAL: NCT03611036
Title: Effect of Different Form of Upper Limb Muscles Training on Dyspnea in COPD
Acronym: REHABSUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REHABSUP (29BRC18.0070)
Record Dates: First submitted 2018-07-16; First posted 2018-08-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength (Experimental): Patients will follow the pulmonary rehabilitation program associated with upper limbs strength training for a duration of 4 weeks
  Interventions: Other: Strength training
- Endurance (Active Comparator): Patients will follow the pulmonary rehabilitation program associated with upper limbs endurance training for a duration of 4 weeks
  Interventions: Other: Endurance training

INTERVENTIONS:
Other: Strength training — Upper limbs Strength training; done with dumbbells whose weight corresponds to 60-80% of the maximal voluntary force in abduction measured initially, during 4 weeks
  Arms: Strength
Other: Endurance training — Upper limbs Endurance training of the ; done with dumbbells whose weight corresponds to 30% of the maximum voluntary force in abduction measured initially, during 4 weeks
  Arms: Endurance

SUMMARY:
Evaluate the effect of upper limbs strength training versus the effect of upper limbs endurance training, on dyspnea, in patients with COPD during a pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patient with stage 2 to 4 (A to D) COPD admitted to a pulmonary rehabilitation program (4 weeks)
* Patient aged 18 or over
* Patient able to consent and having signed a consent form

Exclusion Criteria:

* Patient with pain, osteoarthritis or shoulder surgery
* Patient with a history of Pneumonectomy, lobectomy less than 6 months old
* Refusal of participation
* Patient with an inability to complete a pulmonary rehabilitation program in totality
* Pregnant or breast-feeding women
* Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Compare the effect of upper limbs strength training versus the effect of upper limb endurance training on dyspnea in patients with COPD during a pulmonary rehabilitation program. | Change from inclusion at 4 week
  Measurement of dyspnea using the London Chest Daily Activity Living (LCADL) questionnaire.
  This 15-item, self-administered questionnaire allows an evaluation of dyspnea in patients with COPD during daily activities divided into four components: self-care, domestic, physical, and leisure. Patients could score from 0: "I would not do anyway" to 5: "I need someone else to do this". LCADL score is calculated by aggregating the points assigned to each question, with a higher score representing maximal disability.

SECONDARY OUTCOMES:
Compare dyspnea in daily life between the 2 groups | At inclusion and week 4
  Measurement of dyspnea using mMRC scale. mMRC dyspnea scale is the first self-administered scale which assesses the impact of dyspnea on ADL. It consists of five grades increasing in severity of chronic respiratory disease from 0 : "I only get breathless with strenuous exercise" to 4 : "I am too breathless to leave the house or I am breathless when dressing or undressing."
Compare dyspnea in daily life between the 2 groups | At inclusion and week 4
  Measurement of dyspnea using Dyspnea-12 questionnaire. This 12-item self-administered questionnaire measures dyspnea severity in both its physical and affective components, independently from activity limitation. Patients score ranges from "none" (corresponding to score 0) to "severe" (score 3). Dyspnea-12 score is calculated by aggregating the points assigned to each question; the higher the score, the greater the severity.
Measuring upper limb endurance | At inclusion and week 4
  with the 6-minute Peg Board and Ring Test (6PBRT)
Compare dyspnea at the end of a functional test using the upper limbs | At inclusion and week 4
  Measurement of dyspnea with Borg scale at the end of 6PBRT. The measure is a rating on a scale from 0 to 10 attached to different words of appreciation: "very light, difficult, painful ..." effort.
Compare upper limbs muscle fatigue at the end of a functional test using the upper limbs | At inclusion and week 4
  Measurement of upper limbs muscle fatigue with Borg scale at the end of 6PBRT. The measure is a rating on a scale from 0 to 10 attached to different words of appreciation: "very light, difficult, painful ..." effort.
Compare the evolution of upper limb strength between the 2 groups. | At inclusion and week 4
  Measurement of the strength of deltoids, biceps and brachial triceps, with hand held dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Marc BEAUMONT, PhD, Principal Investigator — CH des pays de Morlaix; Francis COUTURAUD, MD, PhD, Study Director — CHRU de Brest
Locations (2):
- France (2):
  - CHRU de Brest, Brest
  - CH Pays de Morlaix, Morlaix

REFERENCES:
- [Derived] Beaumont M, Peran L, Berriet AC, Ber CL, Courtois-Communier E, Couturaud F. Effect of different forms of upper limb muscle training on dyspnea in chronic obstructive pulmonary disease: a randomised controlled trial. Ann Phys Rehabil Med. 2025 Oct;68(7):102021. doi: 10.1016/j.rehab.2025.102021. Epub 2025 Sep 17. PMID 40966966
- [Derived] Beaumont M, Peran L, Berriet AC, Le Ber C, Le Mevel P, Courtois-Communier E, Couturaud F. Effect of different form of upper limb muscles training on dyspnea in chronic obstructive pulmonary disease: A study protocol. Medicine (Baltimore). 2020 Sep 18;99(38):e22131. doi: 10.1097/MD.0000000000022131. PMID 32957334